CLINICAL TRIAL: NCT00557635
Title: Osseous Setting Improvement With Co-implantation of Osseous Matrix and Mesenchymal Progenitors Cells From Autologous Bone Marrow
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: no recruited patients
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Marc Berger, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0026
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Tibia or Femur Pseudo-arthrosis
Keywords: pseudo-arthrosis, osseous matrix, cell therapy

INTERVENTIONS:
Procedure: Chirurgical procedure — Chirurgical procedure to treat pseudo-arthrosis, with of osseous matrix implantation and autologous bone marrow injection.

SUMMARY:
Sometime osseous reconstruction needs allogeneic bone, in this study we use Ostéopure™ from Ostéobanque d'Auvergne, which is a osseous matrix. However Ostéopure™ integration lasts a long time. To optimize this integration we purpose to associate mesenchymal progenitors cells from autologous bone marrow.

DETAILED DESCRIPTION:
All patients will be treated for tibia or femur pseudo-arthrosis. At the beginning of chirurgical intervention, autologous bone marrow will be sampling and will be concentrated during this one.

Meanwhile osseous matrix (Ostéopure™ ) will be incubated in autologous blood serum and finally implanted in the fracture site. And after (at the end of chirurgical intervention), concentrate autologous bone marrow will be injected in the same place.

ELIGIBILITY:
Inclusion Criteria:

* tibia or femur pseudo-arthrosis,
* patient who needs bone graft

Exclusion Criteria:

* - contra indications for chirurgical intervention or bone graft

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate osseous setting at 3-months follow-up and compare our results with past studies | at 3-months follow-up

SECONDARY OUTCOMES:
Feasibility and tolerance of this therapeutic strategy | at 3-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marc Berger, Dr, Principal Investigator